CLINICAL TRIAL: NCT02197949
Title: Preoperative and Intraoperative Quantification of Axillary Tumoral Load to Reduce the Need of Axillary Lymph Node Dissection in Breast Cancer Patients With Positive Lymph-nodes at Diagnosis
Brief Title: Preoperative and Intraoperative Quantification of Axillary Tumoral Load
Status: Terminated | Type: Observational
Why Stopped: Slow recuitment
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Maria del Mar Vernet, MD, Parc de Salut Mar
Other Study IDs: ELISA
Record Dates: First submitted 2014-07-18; First posted 2014-07-23 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer patients with infiltrated axillary l

SUMMARY:
At present, patients diagnosed of a breast cancer with infiltration of the axillary lymph-nodes are submitted to axillary lymph-node dissection (ALND). The sentinel node (SN) technique is not indicated when a lymph-node biopsy or cytology is positive, nor when the surgical treatment is upfront neither when a neoadjuvant systemic therapy is indicated. The reason for not performing SN is that patients diagnosed of an infiltrated axilla though ultrasound-guided biopsy or cytology tend to have a higher tumoral load than those diagnosed after a sentinel biopsy. Furthermore, even if these patients are submitted to a neoadjuvant systemic treatment and the axillary clinical exploration is negative after the treatment, different studies showed that the SN false negative rate is unacceptably high.

Despite these facts, a high proportion of patients with a positive axilla at diagnosis and submitted to level I and II axillary lymph node dissection show few lymph nodes infiltrated in the pathological study, frequently four or less neoplastic nodes. New methods of detecting these patients with limited infiltrated nodes should be developed and new approaches to axillary surgery (i.e., partial resection) should be offered.

To date, the only information expected to get after an axillary imaging is performed is if the axilla is infiltrated or not. No information about the tumoral load is demanded. In the other hand, level I and II ALND is performed according to established anatomic limits, without selecting the nodes to be excised neither identifying the ones infiltrated for a directed excision.

The aim of the study is to evaluate the ability of a specified and reproducible imaging protocol for distinguishing patients with a high axillary tumoral load from the ones with a low tumoral load. At the same time, as the initial nodes receiving lymph drainage should be the ones commonly affected, identifying these nodes injecting diluted methylene blue in the retroareolar parenchyma and studying their tumoral load could help selecting patients with high from those with low axillary tumoral load.

Evaluation of both steps (that is, first the imaging protocol followed by the methylene blue protocol), could eventually help to distinguish which patients should be submitted to a classical level I and II ALND and which ones can be spared from excising the lymph nodes not stained by the methylene blue.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients with infiltrated axillary lymph nodes cT1-4 cN1
* Older than 18 years old
* Able to understand and accept the protocol procedure and to sign an informed consent form in accordance with national legislation.

Exclusion Criteria:

* Breast cancer patients in whom no information about axillary lymph nodes status (cytology or biopsy) is available.
* Patients younger than 18 years old.
* Psychiatric disease
* Difficulties to understand Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Axillary tumoral load | During surgery (one evaluation)
  -Accuracy to detect patients with low axillary tumoral load (in terms of sensibility and specificity) of a protocol including systematic a reproducible axillary imaging and identification of the first axillary nodes through methylene blue retroareolar injection.

SECONDARY OUTCOMES:
Methylene blue injection to identify nodes of the lymphatic drainage. | During surgery (one evaluation)
  -Identification of clinical data influencing accuracy of methylene blue injection to identify the first four to six lymph nodes of the lymphatic drainage.

CONTACTS AND LOCATIONS:
Overall Officials: Maria del Mar Vernet, MD, PhD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Hospital del Mar, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No